CLINICAL TRIAL: NCT02111980
Title: Compatibility of Radiofrequency Detection Technology With Cardiac Internal Electronic Devices (RF Assure Study)
Brief Title: RF Surgical Sponge-Detecting System on the Function of Pacemakers and Implantable Cardioverter Defibrillators
Acronym: RF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: RF Surgical Systems, Inc. (Industry)
Responsible Party: Principal Investigator, Ulrika Birgersdotter-Green, Professor of Medicine, Cardiac Electrophysiology, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 131198
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Results first posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Cardiomyopathy; Cardiac Arrhythmia; Heart Failure; Chronic Thromboembolic Pulmonary Hypertension
Keywords: CIED; pacemaker; implantable cardioverter defibrillator; ICD; radiofrequency; cardiac device programming; RF sponge detection; RF assure; cardiac internal electronic devices; temporary pacing; pulmonary thromboendarterectomy; pacing interference; Arrhythmia
MeSH Terms: conditions — Cardiomyopathies; Arrhythmias, Cardiac; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RF Assure Scanning (Experimental): The patient's CIED will be interrogated prior to the study to obtain a baseline reading. The patient will be asked to lie down on the RF Assure® Detection Mat with a sponge placed underneath his or her shoulder. The RF Assure® mat and wand will be activated to detect the sponge. The sponge will be removed from underneath the patient's shoulder, and the RF system will be re-activated to obtain a clear reading. The patient's CIED will be re-interrogated to determine if the RF Assure system caused any changes to the CIED parameters or function.
  Interventions: Device: RF Assure Scanning

INTERVENTIONS:
Device: RF Assure Scanning — CIED and temporary pacemaker patients will be scanned with RF surgical sponge detection wand and mat as well as with and without the RF sponge. The scanning will only be conducted on the device scheduled for removal. Patients will have device interrogated before and after scanning (for CIEDs) to determine if there have been any clinically significant changes in programming or settings due to scanning with RF technology. Vitals will be monitored and recorded before, during, and after scanning.

SUMMARY:
If a surgical sponge is mistakenly left inside a patient's body after a surgical procedure, it can cause a serious infection. To prevent this from happening, a new device has been developed that uses radiofrequency (RF) signals to detect the presence of surgical sponges inside the body. The device is now being used routinely to make sure that no sponges are left inside a patient at the end of an operation. However, the RF device has not been implemented in procedures for patients with cardiac implantable electronic devices (CIEDs). While the device is FDA approved for use, there is a theoretical concern that the radiofrequency signals used to detect the sponges will change the settings on the pacemaker or the defibrillator. Changing the settings on a pacemaker might make it pace the heart too quickly or too slowly, while changing the settings on a defibrillator might cause unnecessary shocks or prevent it from shocking the heart if the patient were to have cardiac arrest.

The purpose of this study is to test whether the radiofrequency device used to detect sponges can cause a clinically significant change to the settings on pacemakers and defibrillators. To minimize potential risk, the device will be tested only on patients who are having the pacemaker or defibrillator removed or replaced as part of their regular medical care, either because it is infected or because the battery has worn out. Before the pacemaker or defibrillator is removed, the settings will be carefully and completely recorded and the radiofrequency device will be used to scan the body for sponges as it would be done during normal operation.

After the pacemaker or defibrillator is taken out, the settings will again be recorded and compared to the settings before the scan. In a standard device removal procedure, no clinically significant change in CIED settings would be expected. If a new pacemaker or defibrillator is implanted in the patient, it will not be exposed to the detection device at all. We will also test whether the RF device has any effect on temporary pacemakers that patients may receive after open heart surgery. We plan to perform testing in a total of 50 patients, 40 with permanent pacemakers or defibrillators and 10 with temporary pacemakers.

DETAILED DESCRIPTION:
Retained surgical items (e.g., sponges, needles, and instruments) are among the most frequently reported medical errors and occur in an estimated 1 in 5000 operations. A retained surgical item frequently causes a serious negative outcome, including re-operation (70-80% of cases), readmission or prolonged hospital stay (30-60% of cases), sepsis (43% of cases), or death (2% of cases). Retained surgical items are classed as "never events" by the Centers for Medicare and Medicaid Services (CMS), and CMS does not reimburse for additional medical care related to the treatment for such a complication.

Sponges are by far the most common retained items and are estimated to account for 50-70% of cases. The standard method to ensure that no sponge is left inside the body is manual counting. Manual counting, however, carries a sensitivity and specificity of only about 77% and 99%, respectively. In one study 62% of retained items were detected after the count was reported as normal. If the manual count suggests that a sponge has been retained, the standard method to detect it is by taking a radiograph. Radiographs, however, are time-consuming and in one large retrospective study failed to detect retained items in 33% of cases. The standard methods of detecting retained surgical sponges are clearly suboptimal.

Radiofrequency (RF) technology has recently been employed to improve the detection of retained surgical sponges. A radiofrequency chip is sewn into the fabric of the sponge, and a circular wand that emits a radiofrequency signal is passed over the patient. The wand also serves as an antenna that detects a return signal from the chip in the sponge. If a chip is detected it triggers an audio and a visual alarm on a console attached to the wand. In a study involving 210 patients, RF detection systems had 100% sensitivity and specificity for detecting retained sponges, even in morbidly obese patients. To minimize human error during the scanning process, a new system has been developed where the patient lies on a mat that emits the RF signal and serves as the antenna. In a separate study involving 203 patients, the system using the RF mat had a sensitivity and specificity of 98.5% and 100% respectively. To carry out these studies, sponges were placed underneath patients in a blinded manner. Although it would seem that RF detection systems are superior to manual counting, it should be emphasized that an RF detection system is not a substitute for manual counting, but rather an adjunct to manual counting. The RF Assure ® Detection System manufactured by RF Surgical System Inc. is now routinely used to detect retained sponges in the operating rooms at the University of California, San Diego (UCSD) and at ~200 other hospitals.

There has been some concern that the radio frequency signals emitted by the RF Assure® device might reprogram the settings on CIED such as pacemakers and internal cardiac defibrillators (ICDs), since CIEDs are commonly programmed remotely using RF signals. For this reason, the technology is not commonly used in surgeries with patients with CIEDs. In vitro testing was done in a controlled setting to assess the compatibility of the RF Surgical Detection Technology with permanent pacemakers and ICDs as well as temporary pacemakers, specifically the Boston Scientific Cognis, St. Jude Medical Promote, and Medtronic Virtuoso devices, finding no interference between the RF Assure® system and these devices. Although anecdotal experience and in vitro testing has indicated that the RF Assure® system does not affect CIEDs, it has not been established whether the RF Assure® system is suitable to use in patients with CIEDs in a clinical setting. The purpose of this study is to determine whether the RF Assure® device actually can reprogram CIEDs or cause them to malfunction when used in routine clinical practice. This question is of particular importance because of the rising number of surgical patients, especially cardiac patients, that have an implanted CIED.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age
* Patients must be willing and able to provide consent
* Patients must be eligible for pacemaker/ICD removal or temporary pacemaker

Exclusion Criteria:

* Pregnancy
* Inability or unwillingness to comply with the protocol
* Medical condition that would limit study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika Birgersdotter-Green, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Sulpizio Cardiovascular Center, La Jolla, California, United States

REFERENCES:
- [Background] Cima RR, Kollengode A, Garnatz J, Storsveen A, Weisbrod C, Deschamps C. Incidence and characteristics of potential and actual retained foreign object events in surgical patients. J Am Coll Surg. 2008 Jul;207(1):80-7. doi: 10.1016/j.jamcollsurg.2007.12.047. Epub 2008 May 23. PMID 18589366
- [Background] Egorova NN, Moskowitz A, Gelijns A, Weinberg A, Curty J, Rabin-Fastman B, Kaplan H, Cooper M, Fowler D, Emond JC, Greco G. Managing the prevention of retained surgical instruments: what is the value of counting? Ann Surg. 2008 Jan;247(1):13-8. doi: 10.1097/SLA.0b013e3180f633be. PMID 18156916
- [Background] Gawande AA, Studdert DM, Orav EJ, Brennan TA, Zinner MJ. Risk factors for retained instruments and sponges after surgery. N Engl J Med. 2003 Jan 16;348(3):229-35. doi: 10.1056/NEJMsa021721. PMID 12529464
- [Background] Steelman VM, Alasagheirin MH. Assessment of radiofrequency device sensitivity for the detection of retained surgical sponges in patients with morbid obesity. Arch Surg. 2012 Oct;147(10):955-60. doi: 10.1001/archsurg.2012.1556. PMID 23070411
- [Background] Steelman VM. Sensitivity of detection of radiofrequency surgical sponges: a prospective, cross-over study. Am J Surg. 2011 Feb;201(2):233-7. doi: 10.1016/j.amjsurg.2010.05.001. PMID 21266216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients that required a pacemaker/ICD generator change or device implant were approached for participation in this study in both the Sulpizio Cardiovascular Center Clinic and Pre-procedural Unit. Patients undergoing PTE Surgery were also approached in these settings.
Groups:
- RF Assure Scanning: The patient's CIED was interrogated prior to the study to obtain a baseline reading. The patient was asked to lie down on the RF Assure® Detection Mat with a sponge placed underneath his or her shoulder. The RF Assure® mat and wand were activated to detect the sponge. The sponge was removed, and the RF system was re-activated to obtain a clear reading. The patient's CIED was re-interrogated to determine if the RF Assure system caused any changes to the CIED parameters or function.
  RF Assure Scanning: CIED and temporary pacemaker patients were scanned with RF surgical sponge detection wand and mat as well as with and without the RF sponge. The scanning was be conducted on the device scheduled for removal. Patients had device interrogated before and after scanning (for CIEDs) to determine if there were any clinically significant changes in programming or settings due to scanning with RF technology. Vitals were monitored and recorded before, during, and after scanning.
Period: Overall Study
Arm/Group | RF Assure Scanning
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 50 patients were enrolled in this trial. Of this population, 20 had pacemakers, 20 had ICDs, and 10 were undergoing temporary pacing during Pulmonary Thromboendarterectomy (PTE) surgery.
Groups:
- RF Assure Scanning: Cardiac implantable electronic device (CIED) (implantable cardiac defibrillator (ICD) and permanent pacemakers (PPM)) and temporary pacemaker patients (during pulmonary thromboendartectomy (PTE) surgery) were scanned with the Radiofrequency (RF) surgical sponge detection wand and mat as well as with and without the RF sponge. The scanning was conducted on the device scheduled for removal. Patients had device interrogated before and after scanning (for CIEDs) to determine if there were any clinically significant changes in programming or settings due to scanning with RF technology.
Arm/Group | RF Assure Scanning
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 50 patients were enrolled in this trial. Of this population, 20 had pacemakers, 20 had ICDs, and 10 were undergoing temporary pacing during Pulmonary Thromboendarterectomy (PTE) surgery.
  years
    Pacemaker: number analyzed (Participants) | 20
    Pacemaker | 74.5 (17)
    ICD: number analyzed (Participants) | 20
    ICD | 64 (17.4)
    PTE: number analyzed (Participants) | 10
    PTE | 54.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 50
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: 50 patients were enrolled in this trial. Of this population, 20 had pacemakers, 20 had ICDs, and 10 were undergoing temporary pacing during Pulmonary Thromboendarterectomy (PTE) surgery.
  kg/m^2
    Pacemaker: number analyzed (Participants) | 20
    Pacemaker | 26.3 (3.6)
    ICD: number analyzed (Participants) | 20
    ICD | 29.8 (6.1)
    PTE: number analyzed (Participants) | 10
    PTE | 30.8 (3.9)
History of Coronary Artery Disease (CAD) [Number; unit: participants] — Population: 50 patients were enrolled in this trial. Of this population, 20 had pacemakers, 20 had ICDs, and 10 were undergoing temporary pacing during Pulmonary Thromboendarterectomy (PTE) surgery.
  participants
    Pacemaker: number analyzed (Participants) | 20
    Pacemaker | 6
    ICD: number analyzed (Participants) | 20
    ICD | 6
    PTE: number analyzed (Participants) | 10
    PTE | 1
History of Atrial Fibrillation (AF) [Number; unit: participants] — Population: 50 patients were enrolled in this trial. Of this population, 20 had pacemakers, 20 had ICDs, and 10 were undergoing temporary pacing during Pulmonary Thromboendarterectomy (PTE) surgery.
  participants
    Pacemaker: number analyzed (Participants) | 20
    Pacemaker | 14
    ICD: number analyzed (Participants) | 20
    ICD | 5
    PTE: number analyzed (Participants) | 10
    PTE | 2
History of Diabetes Mellitus (DM) [Number; unit: participants] — Population: 50 patients were enrolled in this trial. Of this population, 20 had pacemakers, 20 had ICDs, and 10 were undergoing temporary pacing during Pulmonary Thromboendarterectomy (PTE) surgery.
  participants
    Pacemaker: number analyzed (Participants) | 20
    Pacemaker | 3
    ICD: number analyzed (Participants) | 20
    ICD | 6
    PTE: number analyzed (Participants) | 10
    PTE | 3
History of Hypertension (HTN) [Number; unit: participants] — Population: 50 patients were enrolled in this trial. Of this population, 20 had pacemakers, 20 had ICDs, and 10 were undergoing temporary pacing during Pulmonary Thromboendarterectomy (PTE) surgery.
  participants
    Pacemaker: number analyzed (Participants) | 20
    Pacemaker | 15
    ICD: number analyzed (Participants) | 20
    ICD | 10
    PTE: number analyzed (Participants) | 10
    PTE | 5
Measured Ejection Fraction (EF) (%) [Mean (Standard Deviation); unit: percentage] — Population: 50 patients were enrolled in this trial. Of this population, 20 had pacemakers, 20 had ICDs, and 10 were undergoing temporary pacing during Pulmonary Thromboendarterectomy (PTE) surgery.
  percentage
    Pacemaker: number analyzed (Participants) | 20
    Pacemaker | 56.2 (17)
    ICD: number analyzed (Participants) | 20
    ICD | 37 (17)
    PTE: number analyzed (Participants) | 10
    PTE | 67.6 (10)

OUTCOME MEASURES:

1. Primary Outcome: Pacing Mode Changes Between Permanent Pacemakers (PPMs)/Implantable Cardiac Defibrillators (ICDs) Scanned With RF Assure
Description: The Pacing Mode on the CIED was measured prior to RF scanning (with sponge) and after the scanning (after sponge removal) in order to evaluate if any significant changes in the pacing mode setting resulted. The following CIED modes were evaluated: DDD (dual chamber pacing, sensing, triggered and inhibited mode), VVI (ventricular pacing, sensing, and inhibited mode), DDI (dual pacing, sensing, and inhibited mode), AAI (atrial pacing, sensing, and inhibited mode). The number of patients' device mode switched between these settings was tabulated and is shown in the below table. Multiple post-scan assessments were not made.
Time Frame: Baseline and 15 minutes
Population: The PTE participants were not included in this analysis because temporary devices do not have capabilities for interrogation (ie: recording pacing mode changes).
Measure: Number; unit: participants
Groups:
- Pre-Scan Measures for PPM/ICDs Scanned With RF Assure: The patient's CIED was interrogated prior to the study to obtain a baseline reading. The patient was asked to lie down on the RF Assure® Detection Mat with a sponge placed underneath his or her shoulder. The RF Assure® mat and wand were activated to detect the sponge. The sponge was removed, and the RF system was re-activated to obtain a clear reading. The patient's CIED was re-interrogated to determine if the RF Assure system caused any changes to the CIED parameters or function.
  RF Assure Scanning: CIED and temporary pacemaker patients were scanned with RF surgical sponge detection wand and mat as well as with and without the RF sponge. The scanning was be conducted on the device scheduled for removal. Patients had device interrogated before and after scanning (for CIEDs) to determine if there were any clinically significant changes in programming or settings due to scanning with RF technology. Vitals were monitored and recorded before, during, and after scanning.
- Post-Scan Measures for PPM/ICDs Scanned With RF Assure: The patient's CIED was interrogated prior to the study to obtain a baseline reading. The patient was asked to lie down on the RF Assure® Detection Mat with a sponge placed underneath his or her shoulder. The RF Assure® mat and wand were activated to detect the sponge. The sponge was removed, and the RF system was re-activated to obtain a clear reading. The patient's CIED was re-interrogated to determine if the RF Assure system caused any changes to the CIED parameters or function.
Arm/Group | Pre-Scan Measures for PPM/ICDs Scanned With RF Assure | Post-Scan Measures for PPM/ICDs Scanned With RF Assure
Number analyzed (Participants) | 40 | 40
participants
  Pacing Mode - DDD | 29 | 29
  Pacing Mode - VVI | 8 | 8
  Pacing Mode - DDI | 2 | 2
  Pacing Mode - AAI | 1 | 1
Statistical Analysis 1: Comparison: Pre-Scan Measures for PPM/ICDs Scanned With RF Assure vs Post-Scan Measures for PPM/ICDs Scanned With RF Assure; Test type: Superiority or Other; p = 1.0, t-test, 2 sided

2. Primary Outcome: Pacing Polarity Changes With Permanent Pacemakers (PPMs)/Implantable Cardiac Defibrillators (ICDs) Scanned With RF Assure
Description: The patient's pacing polarity was measured prior to scanning with sponge and after scanning with sponge via device interrogation. The following pacing polarity measurements were evaluated: right atrium/right ventricle (RA/RV) bipolar polarity, left ventricle (LV) bipolar polarity, and left ventricle (LV) unipolar polarity. Note that not all study patients had LV leads implanted. Multiple post-scan assessments were not made.
Time Frame: Baseline and 15 minutes
Population: The PTE participants were not included in this analysis because temporary devices do not have capabilities for interrogation (ie: recording pacing polarity changes).
Measure: Number; unit: participants
Arm/Group | Pre-Scan Measures for PPM/ICDs Scanned With RF Assure | Post-Scan Measures for PPM/ICDs Scanned With RF Assure
Number analyzed (Participants) | 40 | 40
participants
  RA/RV (bipolar) | 40 | 40
  LV (bipolar) | 5 | 5
  LV (unipolar) | 3 | 3

3. Primary Outcome: Base Rate Measurement Changes With Permanent Pacemakers (PPMs)/Implantable Cardiac Defibrillators (ICDs) Scanned w/ RF Assure
Description: The base rate on patients' devices was measured before scanning with sponge and after RF scanning with sponge. The median was determined and is presented below with standard deviation for both times. Multiple post-scan assessments were not made.
Time Frame: Baseline and 15 minutes
Population: The PTE temporary pacing participants were not included in this analysis because temporary devices do not have capabilities for interrogation (ie: recording base rate measurement changes).
Measure: Median (Standard Deviation); unit: bpm
Arm/Group | Pre-Scan Measures for PPM/ICDs Scanned With RF Assure | Post-Scan Measures for PPM/ICDs Scanned With RF Assure
Number analyzed (Participants) | 40 | 40
bpm | 60 (10.27) | 60 (10.27)

4. Primary Outcome: Max Tracking Rate Changes With Permanent Pacemakers (PPMs)/Implantable Cardiac Defibrillators (ICDs) Scanned With RF Assure
Description: The max tracking rate on the CIEDs was measured prior to scanning with the sponge and post scanning with sponge. The max tracking rate is the maximum atrial rate at which a pacemaker will deliver a ventricular pacing stimulus following each sensed atrial beat. Below, the median and standard deviation are presented. Please note that multiple post-scan assessments were not made for any patient.
Time Frame: Baseline and 15 minutes
Population: 34 of 40 participants' Max Tracking Rate was measured. 6 MTRs were not measured or unable to be measured during testing. The PTE temporary pacing participants were not included in this analysis because temporary devices do not have capabilities for interrogation (ie: recording max tracking rate changes).
Measure: Median (Standard Deviation); unit: bpm
Arm/Group | Pre-Scan Measures for PPM/ICDs Scanned With RF Assure | Post-Scan Measures for PPM/ICDs Scanned With RF Assure
Number analyzed (Participants) | 34 | 34
bpm | 130 (14.51) | 130 (14.51)

5. Primary Outcome: Atrio-ventricular (AV) Delay Changes With Permanent Pacemakers (PPMs)/Implantable Cardiac Defibrillators (ICDs) Scanned With RF Assure
Description: The atrio-ventricular delay was measured prior to scanning with sponge and post RF scanning with sponge. Please note that multiple post-scan assessments were not made for any of the patients presented here.
Time Frame: Baseline and 15 minutes
Population: 31 patients were evaluated of the 40 in this analysis of the AV Delay 9 paced AV Delays were either not measured or unable to be measured during this study. The PTE participants were not included in this analysis because temporary devices do not have capabilities for interrogation (ie: recording AV Delay Changes).
Measure: Median (Standard Deviation); unit: ms
Arm/Group | Pre-Scan Measures for PPM/ICDs Scanned With RF Assure | Post-Scan Measures for PPM/ICDs Scanned With RF Assure
Number analyzed (Participants) | 31 | 31
ms
  Sensed AV Delay | 230 (69.3) | 230 (69.3)
  Paced AV Delay | 250 (68.3) | 250 (68.3)

6. Primary Outcome: Battery Capacity Changes With Permanent Pacemakers (PPMs)/Implantable Cardiac Defibrillators (ICDs) Scanned With RF Assure
Description: Of the patients enrolled, battery capacity changes were measured prior to and post RF scanning with sponge. Multiple post-scan assessments were not made for any of the patients presented here.
Time Frame: Baseline and 15 minutes
Population: Of all participants, only 24 were analyzed in this outcome, as their devices reported battery life in millivolts (while other devices reported battery life in % or years). The PTE temporary pacing participants weren't included in this analysis because temporary devices do not have capabilities for interrogation.
Measure: Median (Standard Deviation); unit: mV
Arm/Group | Pre-Scan Measures for PPM/ICDs Scanned With RF Assure | Post-Scan Measures for PPM/ICDs Scanned With RF Assure
Number analyzed (Participants) | 24 | 24
mV | 2.745 (0.23) | 2.744 (0.23)

7. Primary Outcome: Pacing Impedance Changes With Permanent Pacemakers (PPMs)/Implantable Cardiac Defibrillators (ICDs) Scanned With RF Assure
Description: The impedance values of right ventricle (RV), right atrium (RA), and left ventricle (LV) leads was measured prior to RF scanning with sponge and post RF scanning with sponge. Multiple post-scan assessments were not made for any patient represented here.
Time Frame: Baseline and 15 minutes
Population: 40 subjects were analyzed. Note that not all had both RA, RV, and LV leads. Therefore, the number of leads (and therefore their impedance values reported below) does not match for each group. The PTE temporary pacing participants were not included in this analysis because temporary devices do not have capabilities for interrogation.
Measure: Median (Standard Deviation); unit: ohms
Arm/Group | Pre-Scan Measures for PPM/ICDs Scanned With RF Assure | Post-Scan Measures for PPM/ICDs Scanned With RF Assure
Number analyzed (Participants) | 40 | 40
ohms
  RA Impedance: number analyzed (Participants) | 34 | 34
  RA Impedance | 500.1 (161.18) | 495.1 (161.48)
  RV Impedance: number analyzed (Participants) | 39 | 39
  RV Impedance | 531.9 (135.96) | 530.6 (135.08)
  LV Impedance: number analyzed (Participants) | 8 | 8
  LV Impedance | 592.8 (255.19) | 610.1 (236.89)

8. Primary Outcome: Shock Impedance Changes With Implantable Cardiac Defibrillators (ICDs) Scanned With RF Assure
Description: The shock impedance changes were measured (right ventricle (RV) coil and superior vena cava (SVC) coil) prior to and post RF scanning with sponge. This was measured by performing a device interrogation in the electrophysiology (EP) lab. Multiple post-scan measurements were not taken for any of the patients presented here.
Time Frame: Baseline and 15 minutes
Population: SVC and RV Coils are specific to ICDs, and therefore, PPMs and Temporary Pacemakers were not included in this analysis.
Measure: Mean (Standard Deviation); unit: ohms
Groups:
- Pre-Scan Measures for ICDs Scanned With RF Assure: The patient's CIED was interrogated prior to the study to obtain a baseline reading. The patient was asked to lie down on the RF Assure® Detection Mat with a sponge placed underneath his or her shoulder. The RF Assure® mat and wand were activated to detect the sponge. The sponge was removed, and the RF system was re-activated to obtain a clear reading. The patient's CIED was re-interrogated to determine if the RF Assure system caused any changes to the CIED parameters or function.
  RF Assure Scanning: CIED and temporary pacemaker patients were scanned with RF surgical sponge detection wand and mat as well as with and without the RF sponge. The scanning was be conducted on the device scheduled for removal. Patients had device interrogated before and after scanning (for CIEDs) to determine if there were any clinically significant changes in programming or settings due to scanning with RF technology. Vitals were monitored and recorded before, during, and after scanning.
- Post-Scan Measures for ICDs Scanned With RF Assure: The patient's CIED was interrogated prior to the study to obtain a baseline reading. The patient was asked to lie down on the RF Assure® Detection Mat with a sponge placed underneath his or her shoulder. The RF Assure® mat and wand were activated to detect the sponge. The sponge was removed, and the RF system was re-activated to obtain a clear reading. The patient's CIED was re-interrogated to determine if the RF Assure system caused any changes to the CIED parameters or function.
Arm/Group | Pre-Scan Measures for ICDs Scanned With RF Assure | Post-Scan Measures for ICDs Scanned With RF Assure
Number analyzed (Participants) | 20 | 20
ohms
  RV Coil | 51.30 (18.36) | 51.5 (18.14)
  SVC Coil | 53.45 (17.53) | 53.70 (17.13)

9. Primary Outcome: Changes in P & R Wave Measurements in Permanent Pacemakers (PPMs)/Implantable Cardiac Defibrillators (ICDs) Scanned With RF Assure
Description: The P and R waves were measured via device interrogation prior to and post RF scanning with sponge. Multiple post-scan measurements were not made for any of the participants represented here.
Time Frame: Baseline and 15 minutes
Population: 32 of the 40 participants were evaluated in this study for P and R measurements. 8 patients' devices either didn't have the P or R measured or they was unable to be measured. The PTE temporary pacing participants were not included in this analysis because temporary devices do not have capabilities for interrogation.
Measure: Median (Standard Deviation); unit: mV
Arm/Group | Pre-Scan Measures for PPM/ICDs Scanned With RF Assure | Post-Scan Measures for PPM/ICDs Scanned With RF Assure
Number analyzed (Participants) | 32 | 32
mV
  P Wave | 2.5 (1.38) | 2.469 (1.37)
  R Wave | 10.73 (5.25) | 10.76 (5.29)

10. Primary Outcome: Capture Threshold Changes With Permanent Pacemakers (PPMs)/Implantable Cardiac Defibrillators (ICDs) Scanned With RF Assure
Description: Via device interrogation, capture threshold changes (the minimum amount of electricity that the box has to emit to pace the heart) were measured prior to and post RF Scanning with sponge. Multiple post-scan measurements were not taken for any participants presented here.
Time Frame: Baseline and 15 minutes
Population: Because not all devices are equipped with RA, RV, and LV leads, note the population values in the below table for each group: right atrium (RA) thresholds, right ventricle (RV) thresholds, and left ventricle (LV) thresholds. The PTE participants were not included in this analysis because temporary devices do not have capabilities for interrogation.
Measure: Median (Standard Deviation); unit: V
Arm/Group | Pre-Scan Measures for PPM/ICDs Scanned With RF Assure | Post-Scan Measures for PPM/ICDs Scanned With RF Assure
Number analyzed (Participants) | 40 | 40
V
  RA Threshold: number analyzed (Participants) | 30 | 30
  RA Threshold | 0.806 (0.35) | 0.819 (0.36)
  RV Threshold: number analyzed (Participants) | 39 | 39
  RV Threshold | 0.955 (0.49) | 0.972 (0.50)
  LV Threshold: number analyzed (Participants) | 8 | 8
  LV Threshold | 2.616 (1.16) | 2.320 (1.16)

ADVERSE EVENTS:
Time Frame: Patients were evaluated for adverse events for up to 2 days after their procedure. This was not a follow-up study, therefore, any events that may have occurred after patients were discharged from the hospital were not assessed for this study.
Arm/Group | RF Assure Scanning
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No